CLINICAL TRIAL: NCT06551467
Title: Feasibility Trial of an Innovative Online Ayurveda Program for Detox and Lifestyle: Effect on Mental and Physical Health in Home-Based Adults
Brief Title: Effect of an Innovative Online Ayurveda Program on the Mental and Physical Health of Home-Based Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maharishi International University (Other)
Responsible Party: Principal Investigator, Dr. Viktoria Luhaste, Principal Investigator, Department of Physiology and Health, Maharishi International University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AYU-108-MIU
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Anxiety; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — detox adjuvant

STUDY DESIGN:
Intervention Model Description: This study utilized a single-arm repeated-measures design to monitor changes in the online intervention over time and increase the precision of the outcomes.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): The Online Ayurveda Program for Detox and Lifestyle Intervention Group will be divided into three individual psychophysiological Dosha-specific treatment groups. Participants will be assigned to these groups based on their results from the Ayurveda Dosha Self-Assessment questionnaire.
  Interventions: Behavioral: Online Ayurveda Program for Detox and Lifestyle

INTERVENTIONS:
Behavioral: Online Ayurveda Program for Detox and Lifestyle — The program includes personalized herbal remedies, detoxification procedures, dietary guidelines, yoga exercises, and daily routine practices.

SUMMARY:
The overall objective of this study is to evaluate the effects, feasibility, and safety of a comprehensive online Ayurveda whole-systems (WS) intervention that targets the underlying etiological factors influencing mental and physical health symptoms. The primary hypothesis is that home-based adults who participate in the Ayurveda Program for Detox and Lifestyle will experience a decrease in anxiety and depression symptoms over 4 months.

DETAILED DESCRIPTION:
Two Ayurveda-trained medical doctors will lead the Online Ayurveda Program for Detox and Lifestyle, which comprises eight interactive live webinars over ten days. Each 1.5-hour session includes online group meetings focused on addressing the etiological factors contributing to mental and physical ill-health. The program is easily replicable and includes personalized herbal remedies, detoxification procedures, dietary guidelines, yoga exercises, and daily routine practices, all based on traditional Ayurvedic medicine principles. After the ten-day detoxification, participants will continue to follow the diet and lifestyle recommendations and the herbal program for mental and physical health for up to four months. Outcome measures will be assessed at baseline and once a month for four months.

ELIGIBILITY:
Inclusion Criteria:

* Scored ≥ 5 on the GAD-7
* Scored ≥ 5 on the PHQ-9
* Scored ≥ 5 on the PHQ-15
* Age 18-80 years
* No other psychiatric disorders
* Not receiving specialized treatments for anxiety or depression, nor participating in another clinical trial
* Stable psychiatric medication regimen for more than two months
* No acute or severe medical conditions
* Individuals who are not pregnant or breastfeeding
* Provided informed consent

Exclusion Criteria:

* Scored < 5 on the GAD-7
* Scored < 5 on the PHQ-9
* Scored < 5 on the PHQ-15
* Age under 18 or over 80 years
* Other psychiatric disorders (e.g., suicidal risk)
* Currently undergoing specialized treatments for anxiety and depression, or participating in another clinical trial
* Psychiatric medication regimen for less than 2 months
* Acute or severe medical condition (e.g., stroke, surgery)
* Individuals who are pregnant or breastfeeding
* Inability to provide informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2022-07-25 (Actual)

PRIMARY OUTCOMES:
Change in Anxiety Score | Assessed at baseline and once a month for four months
  Assessed using the online standardized Patient Health Questionnaire for Somatic, Anxiety, and Depressive Symptoms (PHQ-SADS). The PHQ-SADS uses cut-off points of 5, 10, and 15 to represent mild, moderate, and severe symptoms, respectively. The assessment includes the Generalized Anxiety Disorder 7-item (GAD-7) scale, which measures the severity of anxiety. The GAD-7 uses cut-off points of 5, 10, and 15 for mild, moderate, and severe anxiety, respectively. The scale ranges from 0 to 21, with higher scores indicating greater anxiety levels.
Change in Depression Score | Assessed at baseline and once a month for four months
  Assessed using the online standardized Patient Health Questionnaire for Somatic, Anxiety, and Depressive Symptoms (PHQ-SADS). The PHQ-SADS uses cut-off points of 5, 10, and 15 to represent mild, moderate, and severe symptoms, respectively. The assessment also includes the Patient Health Questionnaire-9 (PHQ-9) for depression, which uses cut-off points of 5, 10, 15, and 20 to represent mild, moderate, moderately severe, and severe depression, respectively. The PHQ-9 scale ranges from 0 to 27, with higher scores indicating greater severity of depression.

SECONDARY OUTCOMES:
Change in Somatic or Physical Symptoms Score Change in Somatic or Physical Symptoms Score | Assessed at baseline and once a month for four months
  Assessed using the online standardized Patient Health Questionnaire for Somatic, Anxiety, and Depressive Symptoms (PHQ-SADS). The PHQ-SADS uses cut-off points of 5, 10, and 15 to represent mild, moderate, and severe symptoms, respectively.
  The assessment also includes the PHQ-15 scale, which assesses somatic symptoms. The PHQ-15 uses cut-off points of 5, 10, and 15 to represent mild, moderate, and severe somatic symptoms, respectively. The scale ranges from 0 to 30, with higher scores indicating greater severity of somatic symptoms.
Change in Fatigue Score | Assessed at baseline and once a month for four months
  Fatigue was measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue Short Form (8a). The form uses a scale of 8 to 40, with higher scores indicating more significant fatigue. Scores of 22, 26, and 36 represent mild, moderate, and severe fatigue.
Changes in Body Mass Index (BMI) | Assessed at baseline and once a month for four months
  Participants measured their height and weight using a standard scale and tape, and then reported these measurements in the online survey. Body Mass Index (BMI) was calculated using the standardized formula: weight (kg) / [height (m)]². The calculations were performed using an Excel program.

CONTACTS AND LOCATIONS:
Overall Officials: Viktoria Luhaste, PhD, Principal Investigator — Maharishi International University
Locations (1):
- The Center for Maharishi AyurVeda and Holistic Medicine, Geboltskirchen, Austria

IPD SHARING:
Plan to Share IPD: Yes
The research data supporting this study's findings are not publicly accessible due to privacy and ethical constraints related to patient consent. However, anonymized data may be available from the authors upon request with permission from the institutional review board of Maharishi International University, Fairfield, Iowa.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be available six months after the study results are published in a peer-reviewed journal and will be accessible for up to three years after that.
Access Criteria: Researchers must submit a methodologically sound proposal for review by the data-sharing committee and the institutional review board of Maharishi International University, Fairfield, Iowa. The committee will approve access, and a data use agreement must be signed prior to data release.